CLINICAL TRIAL: NCT04389736
Title: Effects of Self-selected Maiximal Intensity of Neuromuscular Electrical Stimulation (NMES) on Energy Expenditure, Glycaemia and Hormonal Responses on Healthy Individuals
Brief Title: Effects of NMES on Energy Expenditure, Glycaemia and Hormonal Responses to Glucose Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Collaborators: University of Bath (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EP 17/18 230
Record Dates: First submitted 2020-03-27; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Energy Expenditure; Metabolic Health
Keywords: Neuromuscular electrical stimulation; Insulin resistance; Standing; Glucose control
MeSH Terms: conditions — Insulin Resistance | interventions — Sitting Position; Standing Position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SIT (Experimental): Sitting
  Interventions: Behavioral: Sitting
- STAND (Experimental): Standing
  Interventions: Behavioral: Standing
- NMES (Experimental): Self-selected maximal intensity of neuromuscular electrical stimulation
  Interventions: Behavioral: Self-selected maximal intensity of neuromuscular electrical stimulation

INTERVENTIONS:
Behavioral: Sitting — Participants sat in a chair with back, arms and legs supported.
  Arms: SIT
Behavioral: Standing — Participants were asked to stand with arms supported and feet spaced approximately 15 cm apart. If needed, adjustment of standing posture was allowed during standing trial to prevent orthostatic hypotension.
  Arms: STAND
Behavioral: Self-selected maximal intensity of neuromuscular electrical stimulation — Small electrodes placed (5*5 cm) on the lower limb of both legs. The instruction for NMES intensity was that the maximal intensity participants were be able to withstand for 2 hours whilst imagining sitting at home watching TV without feeling discomfort.
  Arms: NMES

SUMMARY:
The purpose of this study is to investigate whether self-selected neuromuscular stimulation (NMES) affects energy expenditure, glycaemia and hormonal responses in healthy men and women

DETAILED DESCRIPTION:
Participants were asked to perform 3 trials [sitting (SIT), standing (STAND) and sitting with neuromuscular electrical stimulation (NMES) to the lower limbs in randomised counter-balanced study design. Trials were separated by at least 48 h and were completed within 14 days. In all trials, participants were required to remain relaxed and motionless. SIT: participants sat in a chair with back, arms and legs supported. STAND: participants were asked to stand with arms supported and feet spaced approximately 15 cm apart. If needed, adjustment of standing posture was allowed during the standing trial to prevent orthostatic hypotension. NMES: prior to the NMES trial, participants underwent preliminary testing to ensure that stimulation was comfortable. Before the NMES, a small area of the body hair was shaved and skin was cleaned with an alcohol wipe and electrodes were stuck to the surface of the skin. Small electrodes placed (5*5 cm) on the lower limb of both legs (gastrocnemius, rectus femoris, vastus medialis). The two devices (EM 80, Beurer UK Ltd, Golborne, UK) were set up with the frequency of 20 Hz along with stimulation period of 1 second on and 1 second off throughout a 2 h oral glucose tolerance test (OGTT). The instruction for NMES intensity was that the maximal intensity participants were be able to withstand for 2 hours whilst imagining sitting at home watching TV without feeling discomfort. Prior to the OGTT, 5 min was given to identify the suitable intensity of stimulation and within the first 10 min of the OGTT participants were allowed to adjust the intensity once, after which, the intensity remained the same for the rest of OGTT. Participants were asked to sit in a chair with back, arms and legs supported during the stimulation. During trials, participants could watch TV, or read, but typing on a laptop or computer were avoided.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Aged between 18 to 65 years
* Weight stable for more than 3 months (no change in weight +/- 3%)
* Non-smoker

Exclusion Criteria:

* Personal history of/existing diabetes, cardiovascular disease, metabolic disease or dyslipidaemia
* Taking medications that may influence lipid or carbohydrate metabolism or immune system function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Changes in total energy expenditure during OGTT test. | 120 minutes
  Changes in total energy expenditure during OGTT test.

SECONDARY OUTCOMES:
Changes in blood glycaemic responses during OGTT test. | 120 minutes
  Changes in blood glycaemic responses during OGTT test.
Changes in blood insulinaemic responses during OGTT test. | 120 minutes
  Changes in blood insulinaemic responses during OGTT test.
Changes in blood pressure during OGTT test. | 120 minutes
  Changes in blood pressure during OGTT test.
Changes in heart rate during OGTT test. | 120 minutes
  Changes in heart rate during OGTT test.
Changes in gut hormones (GLP-1, GIP & PYY etc.) responses during OGTT test. | 120 minutes
  Changes in gut hormones (GLP-1, GIP & PYY etc.) responses during OGTT test.
Changes in total carbohydrate during OGTT test. | 120 minutes
  Changes in total carbohydrate during OGTT test.
Changes in total lipid oxidation during OGTT test. | 120 minutes
  Changes in total lipid oxidation during OGTT test.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

REFERENCES:
- [Derived] Chen Y.-C., Davies R.G., Hengist A., Carroll H.A., Perkin O.J., Betts J.A., Thompson D.. Effects of neuromuscular electrical stimulation on energy expenditure and postprandial metabolism in healthy men. Appl Physiol Nutr Metab. 2022 Jan;47(1):27-33. doi: 10.1139/apnm-2021-0361. Epub 2021 Aug 17. PMID 34403626